CLINICAL TRIAL: NCT05828121
Title: Preventing an Opioid Epidemic in Norway: Focusing on Treatment of Chronic Pain
Brief Title: POINT - Preventing an Opioid Epidemic in Norway: Focusing on Treatment of Chronic Pain
Acronym: POINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kine Gjesdal, Associate professor, Helse Stavanger HF
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: POINTstavanger
Record Dates: First submitted 2023-02-08; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain; Opioid Use
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: MRC framework for a complex intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Point1 (Experimental): Receiving treatment
  Interventions: Behavioral: POINT1

INTERVENTIONS:
Behavioral: POINT1 — Receiving treatment

SUMMARY:
The investigators do research on chronic pain treatment to minimize the risks associated with opioids.

DETAILED DESCRIPTION:
The investigators know that patients suffering from chronic pain need good treatment. The use of opioids for chronic, non-cancer related pain may seem appropriate in the short term, but can often have negative consequences for both the individual and society in the long term.

Several factors-the escalating use of opioids to chronic pain patients, the increasing use of strong opioids in particular, and the increasing number of overdoses caused by prescription opioids-point to the start of an opioid epidemic in Norway.

Objectives The overall goal of the POINT project is to provide knowledge to optimize treatment of patients with chronic pain in order to avoid unnecessary escalation of opioid treatment, improve their quality of life and reduce the burden of disease.

In the long run our objective is to prevent the unwanted consequences of opioid treatment and improve patients' quality of life.

Ultimately, through this project the investigators hope to prevent an opioid epidemic in Norway.

To achieve the main goal, the investigators will focus on pain patients and their doctors, as increasing opioid use may occur through the patient-doctor interaction.

Methods

The project will develop and test a non-drug interventions that consist of an interdisciplinary group treatment .

Financing The Research Council of Norway

Cooperation St. Olavs Hospital

Stavanger Hospital Trust

City of Stavanger

National Institute of Public Health (FHI)

Alcohol and Drug Research Western Norway (KoRFor)

Foreningen for kroniske smertepasienter (FKS) Norwegian Forum of Disabled Peoples' Organizations (SAFO)

Cooperation with other projects Injury Prevention and Outcomes following Trauma

ELIGIBILITY:
Inclusion Criteria:

* non-malignant, chronic pain
* Registered in Stavanger municipality
* Consent to participation.
* Age 18 - 67 years
* Pain duration <10 years

Exclusion Criteria:

* malignant pain condition

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Audit C at 12 Weeks | 12 weeks
  Audit C
Change from baseline in Pain Scores on the Visual Analog Scale at 12 Weeks | 12 weeks
  Visual Analog Scale
Change from baseline in Bergen Insomnia scale at 12 Weeks | 12 weeks
  BIS
Change from baseline in Health-related quality of life at 12 Weeks | 12 weeks
  HQ5D5L

CONTACTS AND LOCATIONS:
Locations (1):
- Stavanger municipality, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2023